CLINICAL TRIAL: NCT02085876
Title: Quantitative and Qualitative MRI Study of Steatosis in Patients With Metabolic Steatopathy
Acronym: IRM Stéatose
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: HAMZA APJ 2013
Record Dates: First submitted 2014-03-05; First posted 2014-03-13 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2013-07

CONDITIONS: Overweight; Type 2 Diabetes; Obesity
Keywords: patients; present; undergo bariatric surgery
MeSH Terms: conditions — Overweight; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients requiring a liver biopsy
  Interventions: Other: 2 additional MRI sequences; Other: An additional blood sample

INTERVENTIONS:
Other: 2 additional MRI sequences
Other: An additional blood sample

SUMMARY:
This is a single centre prospective open-label, non-randomised pilot study whose aim is to identify MRI parameters to better evaluate inflammation and liver fibrosis and thus, in the near future, to avoid the need for liver biopsy.

To achieve this:

* The MRI study will be completed by adding two sequences: Measurement of T1 and multiecho T2*. The other data will be extracted from usual sequences.
* Part of the histological samples will be used for the weighted levels of fat and iron, and for the lipidomic study.
* Usual blood samples will be completed by samples for the serum library

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been informed about the research
* Patients with national health insurance cover
* Patients who are overweight (BMI > 25) or have type 2 diabetes suggesting a disturbance of hepatic enzymes (ASAT < 8 times normal values and ALAT > twice normal values) after a complete hepatopathy assessment
* Obese patients with a hepatic anomaly (steatosis) revealed by imaging or biological assessment (ASAT < 8 times normal values and ALAT > twice normal values) who are eligible for bariatric surgery and a preoperative liver MRI examination.

Exclusion Criteria:

* Non-corrected coagulation disorder.
* Patients aged over 80 years
* Patients aged less than 18 years
* Patients without legal protection
* Patients with a contra-indication for MRI (Pacemaker, intraocular metallic foreign body, weight>150kg)
* Patients without national health insurance cover

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Overweight patients or patients with type 2 diabetes or obese patients (who present a liver anomaly and should undergo bariatric surgery)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Primary Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
To determine a correlation coefficient > 0.80, alpha 0.05 and beta 0.20 between the MRI markers relevant. | Baselines

SECONDARY OUTCOMES:
To determine the correlation between the unsaturated fat measurements and MRI Lipidomics Spectro analysis. | Baselines

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France